CLINICAL TRIAL: NCT06658301
Title: Comparative Study on the Effectiveness of Plyometric Push up and Swiss Ball Push up in the Management of Throwing Distance and Accuracy Among Badminton Players
Brief Title: Comparative Study on the Effectiveness of Plyometric PU and Swiss Ball PU in Badminton Players
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0427
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Sports Physical Therapy
Keywords: Agility; Plyometric exercise; Strenght

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plyometric push up exercises (Experimental): The subjects will starts with push-up position with hands on the floor, place slightly wider than shoulder width apart and their feet together. Keeping their back flat, slowly lower the body toward the ground. Then in one explosive movement, push-up and away from the floor as quickly as possible, bring their hands off the floor.
  Interventions: Other: plyometric push up exercises
- swiss ball push up exercises (Experimental): The subjects will start with kneeling position so that they will face the ball. Place their hands on top of the ball so that they can bend their elbows towards the body. Straight the legs out and raise themselves slightly higher so that they can be on their toes. Stay in neutral position. Straighten their arms at the elbows, so that they can push themselves up from the ball.
  Interventions: Other: swiss ball push up exercises

INTERVENTIONS:
Other: plyometric push up exercises — The subjects will starts with push-up position with hands on the floor, place slightly wider than shoulder width apart and their feet together. Keeping their back flat, slowly lower the body toward the ground. Then in one explosive movement, push-up and away from the floor as quickly as possible, bring their hands off the floor.
  Arms: plyometric push up exercises
Other: swiss ball push up exercises — . The subjects will start with kneeling position so that they will face the ball. Place their hands on top of the ball so that they can bend their elbows towards the body. Straight the legs out and raise themselves slightly higher so that they can be on their toes. Stay in neutral position. Straighten their arms at the elbows, so that they can push themselves up from the ball.
  Arms: swiss ball push up exercises

SUMMARY:
The aim of this study is to find out the comparative effect of plyometric push up and swiss ball push up in the management of throwing distance and accuracy among badminton player.

DETAILED DESCRIPTION:
In previous researches, little literature is available regarding comparison of the effectiveness of plyometric push-up and Swiss ball push-up specifically in the management of throwing distance in badminton players. There is a dire need to explore the comparative effects of these two training methods within the context of badminton. Moreover, Further studies exploring different approaches for throwing accuracy in badminton players are required in the existing researches.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and Females
* Age 16-30 years
* Sporting activity of minimum 40 minutes thrice a week
* Subjects being engaged in sports that require athlete's arm to be above shoulder height on a repetitive basis during throwing.

Exclusion Criteria:

* Spinal deformity
* Cervical spine pathology
* Glenohumeral subluxation
* Any recent upper limb fracture
* Recent Rotator cuff tear
* Bone disease
* Glenohumeral dislocation

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Functional throwing performance index | 6 weeks
  Functional ability of the shoulder joint will be assessed using FTPI. The subject stood 15ft from a target, a 1ftx1ft square on at a height of 4ft from the floor. The object of the test is to throw a standard leather ball into the target as many times as possible over 30 second trails. Before testing, subject's will perform 8 throws as a warm-up. Test began immediately after the warm-up consists of the subject 22 throwing the ball into the target, catching the rebound of the wall and repeating as many times as possible within 30 seconds. The FTPI is calculated as the number throws with in the target divided by total number of balls thrown.
Medicine ball throw test | 6 weeks
  Medicine ball throw test will be used to assess upper-body explosive power. Throwing distance will be measured by using the medicine ball throw test. In this test, participants will be instructed to throw a medicine ball as far as they could, in a walk stand position, holding the ball overhead with the dominant hand. The medicine ball will be used had a mass of 2 kg and diameter 56cm each subject performed 5 trials with 1 min rest between trails. The distance in meter to which the subject threw the medicine ball was measured with the measuring tape. The best of 5 trials will be taken and used for further analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Rikza Khalid, DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ikeda Y, Kijima K, Kawabata K, Fuchimoto T, Ito A. Relationship between side medicine-ball throw performance and physical ability for male and female athletes. Eur J Appl Physiol. 2007 Jan;99(1):47-55. doi: 10.1007/s00421-006-0316-4. Epub 2006 Oct 18. PMID 17047981
- [Background] Bodden D, Suchomel TJ, Lates A, Anagnost N, Moran MF, Taber CB. Acute Effects of Ballistic and Non-ballistic Bench Press on Plyometric Push-up Performance. Sports (Basel). 2019 Feb 18;7(2):47. doi: 10.3390/sports7020047. PMID 30781654
- [Background] Pisz A, Blazek D, Jebavy R, Kolinger D, Wilk M, Krzysztofik M, Stastny P. Antagonist activation exercises elicit similar post-activation performance enhancement as agonist activities on throwing performance. BMC Sports Sci Med Rehabil. 2023 Mar 27;15(1):44. doi: 10.1186/s13102-023-00657-9. PMID 36973790
- [Background] Arakaki JS, Jennings F, Estrela GQ, Cruz Martinelli VDG, Natour J. Strengthening exercises using swiss ball improve pain, health status, quality of life and muscle strength in patients with fibromyalgia: a randomized controlled trial. Reumatismo. 2021 Apr 19;73(1):15-23. doi: 10.4081/reumatismo.2021.1357. PMID 33874643
- [Background] Zubac D, Paravlic A, Koren K, Felicita U, Simunic B. Plyometric exercise improves jumping performance and skeletal muscle contractile properties in seniors. J Musculoskelet Neuronal Interact. 2019 Mar 1;19(1):38-49. PMID 30839302
- [Background] Van Roie E, Walker S, Van Driessche S, Delabastita T, Vanwanseele B, Delecluse C. An age-adapted plyometric exercise program improves dynamic strength, jump performance and functional capacity in older men either similarly or more than traditional resistance training. PLoS One. 2020 Aug 25;15(8):e0237921. doi: 10.1371/journal.pone.0237921. eCollection 2020. PMID 32841300
- [Background] Sha Z, Dai B. The validity of using one force platform to quantify whole-body forces, velocities, and power during a plyometric push-up. BMC Sports Sci Med Rehabil. 2021 Aug 30;13(1):103. doi: 10.1186/s13102-021-00330-z. PMID 34462003
- [Background] Bezerra ES, Orssatto LBDR, Werlang LC, Generoso AM, Moraes G, Sakugawa RL. Effect of push-up variations performed with Swiss ball on muscle electromyographic amplitude in trained men: A cross-sectional study. J Bodyw Mov Ther. 2020 Apr;24(2):74-78. doi: 10.1016/j.jbmt.2019.09.004. Epub 2019 Sep 10. PMID 32507156
- [Background] Kossow AJ, Ebben WP. Kinetic Analysis of Horizontal Plyometric Exercise Intensity. J Strength Cond Res. 2018 May;32(5):1222-1229. doi: 10.1519/JSC.0000000000002096. PMID 29533358
- [Background] Dhahbi W, Chaabene H, Chaouachi A, Padulo J, G Behm D, Cochrane J, Burnett A, Chamari K. Kinetic analysis of push-up exercises: a systematic review with practical recommendations. Sports Biomech. 2022 Jan;21(1):1-40. doi: 10.1080/14763141.2018.1512149. Epub 2018 Oct 4. PMID 30284496
- [Background] Zalleg D, Ben Dhahbi A, Dhahbi W, Sellami M, Padulo J, Souaifi M, Beslija T, Chamari K. Explosive Push-ups: From Popular Simple Exercises to Valid Tests for Upper-Body Power. J Strength Cond Res. 2020 Oct;34(10):2877-2885. doi: 10.1519/JSC.0000000000002774. PMID 30095736
- [Background] Malwanage KT, Senadheera VV, Dassanayake TL. Effect of balance training on footwork performance in badminton: An interventional study. PLoS One. 2022 Nov 17;17(11):e0277775. doi: 10.1371/journal.pone.0277775. eCollection 2022. PMID 36395192
- [Background] Falch HN, Raedergard HG, van den Tillaar R. Association of strength and plyometric exercises with change of direction performances. PLoS One. 2020 Sep 10;15(9):e0238580. doi: 10.1371/journal.pone.0238580. eCollection 2020. PMID 32911530